CLINICAL TRIAL: NCT03432572
Title: Pilot Study: Investigating Oral Agents for Urine Staining to Facilitate Intraoperative Observation of Ureteral Jets
Brief Title: Investigating Oral Agents for Urine Staining to Facilitate Intraoperative Observation of Ureteral Jets
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: L18-072
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Ureteral Injury
MeSH Terms: interventions — Phenazopyridine; Riboflavin; Thiamine

STUDY DESIGN:
Intervention Model Description: This will be a 3 arm randomized controlled double blinded study. The arms will all be studied in parallel to each other and compared in their effectiveness for evaluation for urine jets on cystoscopy.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The interventions will be blinded to the investigator, the care providers (surgeons), and will be blinded to the patients in the study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- pyridium (Experimental): Group A will take 200 mg of oral Pyridium 1 hour before surgery and then the urine jets will be evaluated on cystoscopy in the operating room during a gynecological procedure.
  Interventions: Drug: Pyridium
- riboflavin (Active Comparator): Group B will take 400 mg of riboflavin 1 hour before surgery and then the urine jets will be evaluated on cystoscopy in the operating room during a gynecological procedure.
  Interventions: Drug: Riboflavin
- thiamine (Placebo Comparator): Group C will take the placebo (50 mg of thiamine) 1 hour before surgery and then the urine jets will be evaluated on cystoscopy in the operating room during a gynecological procedure.
  Interventions: Drug: Thiamine

INTERVENTIONS:
Drug: Pyridium — a urine discoloration agent
  Other Names: Group A
  Arms: pyridium
Drug: Riboflavin — a urine discoloration agent
  Other Names: Group B
  Arms: riboflavin
Drug: Thiamine — active placebo not known to cause urine discoloration
  Other Names: Group C
  Arms: thiamine

SUMMARY:
Recently, Indigo Carmine and Methylene Blue have been the standard agents to visualize ureteral jets during intraoperative cystoscopy. However, due to a national shortage of Indigo Carmine and Methylene Blue, there is a need to discover alternative IV and oral agents that are readily available and well tolerated when used for visualizing ureteral jets at the time of intraoperative cystoscopy. The aim of this study is to look at oral agents that have been studied such as pyridium (Phenazopyridine Hydrochloride) and riboflavin and compare them in a three-arm double-blinded randomized controlled pilot study using riboflavin, pyridium, and a placebo. The aim of the study is to provide evidence that both pyridium and riboflavin are effective and safe for staining urine to facilitate visualization of jets in evaluating ureteral patency at the time of intraoperative cystoscopy.

DETAILED DESCRIPTION:
This is a 3 arm, double- blinded, randomized, controlled pilot study to look at the ease of evaluating ureteral patency at the time of intraoperative cystoscopy and comparing effects and possible adverse effects of these two interventions compared to subjects receiving a placebo. The interventions will be blinded to the investigators and to the participants. The Clinical Research Institute in the Texas Tech Health Sciences Center will assist with randomization techniques for administering the agents to the subjects. The subjects will take the agents on the morning of surgery 1 hour (+/- 15 minutes) prior to the procedure.

Group A will take 200 mg of oral Pyridium 1 hour before surgery. Group B will take 400 mg of riboflavin 1 hour before surgery. The placebo, 50 mg of vitamin B1 thiamine, will be administered to Group C patients. Group C will take the placebo (50 mg of thiamine) 1 hour before surgery. This study will be double blinded. There will be a third party who prepares an envelope for the patient. The patient will be unaware of which one it will be, but will have appropriate consent ahead of time. The physicians doing the case will be blinded to which agent was administered to the patient. A data collection sheet will be filled in by a member of the study team. Body Mass Index (BMI), height, weight, Liver Function Tests (LFTs), creatinine, and time from ingestion to time of cystoscopy will be recorded. Additionally, the surgeons will complete a survey regarding the stain of the urine and quality of the urine jet. The investigators will have the options of writing in no color, slightly colored, or bright colored urine and for the jet the investigators will have the options of trickle, moderate jet, or strong jet. These data will be collected and then entered into a database and analyzed for statistical significance. In this study, the investigators will define statistical significance as an alpha value of < 0.05 with respect to the riboflavin and pyridium study groups compared with the control group. The data collection sheet represents a semi-quantitative color and flow grading system.

Randomization will occur just prior to surgery. A randomization list will be generated by the statisticians in the Clinical Research Institute (CRI). Randomization will be through a series of sealed envelopes containing equal numbers of Group A, Group B and Group C allocations. Following enrollment, the study coordinator will draw the next sequential numbered envelope and proceed according to group assignment. A master list will be kept of patient identification (ID) and randomization assignment by an independent third party.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 75 years.
2. Female patients ages who are scheduled to undergo gynecologic procedures where cystoscopy/need to determine ureteral patency may be indicated.
3. Being seen in the department of Texas Tech OB/GYN.
4. Willing to be randomized.
5. Have not taken, or willing to stop taking pyridium or riboflavin at least 7 days prior to surgery.

Exclusion Criteria:

1. Female patients who are found to have one of the following conditions based on their medical history: Active Inflammation of the Liver, Glomerulonephritis, Uremia, Kidney Disease, Glucose-6-Phosphate Dehydrogenase (G6PD) Deficiency, Anemia from Pyruvate Kinase and G6PD Deficiency.
2. Patients who have allergies to pyridium, riboflavin, or vitamin B1 riboflavin.
3. Patients who, for whatever reason, did not receive the product they were randomized to receive.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
urine discoloration on cystoscopy | through study completion, an average of 1 year
  To determine if oral pyridium and vitamin B riboflavin administration prior to gynecologic procedures are effective and safe alternatives for evaluating ureteral patency at the time of cystoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia DeRiese, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States